**Study Code:** NOV2019/01864 NCT04639869 **Date:** 13.05.2019 **Version:** 1.0

Subject Screening Number: .....

## INFORMED CONSENT FORM

Principal Investigator: Prof. Dr. Muradiye Nacak

Gaziantep Üniversitesi FARMAGEN GCP Center

Gaziantep Üniversitesi Teknoloji Geliştirme Bölgesi (Teknopark)

Burç Yolu, Şahinbey 27260, Gaziantep-Turkey

Telephone: +90 342 360 62 62 GSM: +90 505 252 54 69

"Open-label, randomised, single oral dose, four-period, replicated, cross-over trial to assess the bioequivalence of Feniramidol HCl 400 mg Film Tablet (Test Drug) in comparison with Cabral 400 mg Film Tablet (Reference Drug) in healthy male subjects under fed conditions"

## Dear Volunteer,

The drug tested in this trial is Feniramidol HCl 400 mg Film Tablet, containing 400 mg phenyramidol hydrochloride of Pharmactive İlaç San.ve Tic. A.Ş. It is a medication used orally and it could be valuable in the treatment of painful muscle spasms.

The purpose of the present research study is to investigate the bioequivalence of orally administered test drug containing 400 mg phenyramidol hydrochloride (Feniramidol HCl 400 mg Film Tablet) and on the other orally administered reference drug containing 400 mg phenyramidol hydrochloride (Cabral 400 mg Film Tablet). The reference drug is already registered and commercially available for years in Turkey as Cabral 400 mg Film Tablet. The company responsible for placing the reference product on the market is Recordati İlaç San. ve Tic. A.Ş., Turkey. The efficacy and safety of this reference drug has been proven through the clinical studies that were carried out in order to obtain the license for the drug. Therefore, this drug will be used as reference and will establish the basis of comparison to be used for the test drug (Feniramidol HCl 400 mg Film Tablet). (Feniramidol HCl 400 mg Film Tablet is manufactured by Pharmactive İlaç San.ve Tic. A.Ş. in Turkey.) The comparison will be based on the measurement of the concentrations of the active ingredient of the drugs in blood. In addition, the safety of the test product will be compared to the safety of the reference products based on the evaluation of adverse events.

Under fed condition in this 4 period trial, each of 44 subjects who enrolled into trial will be given a single dose of the test (T) or the reference (R) drug orally (Test Drug or Reference Drug= single dose of 400 mg phenyramidol hydrochloride in each period) and there will be a wash-out of at least 7 days. You will take a total of 1600 mg phenyramidol hydrochloride during the trial. The drugs will be assigned randomly. Therefore, you will have an equal chance of receiving either drug. The total duration of the trial will be approximately 6 weeks.

Screening tests will be done before the beginning of the study and will include standard clinical and laboratory research lasting no more than 14 days. Standard clinical research includes your medical history, a complete clinical examination, drug abuse screening, alcohol breath test, standard ECG, and measurement of your height, weight, body temperature, blood pressure, and heart rate after five minutes of rest in the supine position.

The final examination will be carried out on the day of last blood sampling in the last period or not more than 7 days thereafter and will include standard clinical and laboratory research. Standard clinical research includes a complete clinical examination, standard ECG, body temperature, blood pressure, and heart rate after five minutes of rest in the supine position.

Approximately 32 mL blood sample (20\* mL for entry examination and 12 mL for final examination) is going to be collected for the standard laboratory tests on entry and final examination with HIV (AIDS) and hepatitis tests at only entry examination. The blood samples collected for laboratory (entry and final examination) tests will be sent to GAMA Medical Laboratories (GAMA Tip Laboratuvarlari) which is located in Gaziantep-Turkey, and will be used exclusively for this research, specifically for it's purpose. An amount of blood sample will be needed if any Clinical Laboratory Tests occur which need to be repeated.

\* 8 mL of 20 mL of entry examination blood sample will be used for analytical studies of this project.

Approximately 30 mL urine sample is going to be collected for the standard laboratory tests on entry and final examination with drug abuse tests on entry examination and day 0 (hospitalization/randomisation day) of each period.

You will come to the clinic the day before each drug administration period around 18:00 and will stay in the clinic until 10 hours after the drug is given. But according to your health situation, the investigator and/or co-investigator will be decided whether you can leave the clinic at that time or not. Your body temperature will be measured in the evening before the administration of the drug in each period. You will have to come to the clinic for a final examination and laboratory tests on the day of last blood sampling in the 4<sup>th</sup> period or not more than 7 days thereafter.

You should not consume alcohol and cigarette during the trial. You will not be allowed to chewing gum on the day of drug administration. You will not be allowed to consume food or drink (coffee, tea, cola, hot chocolate, etc.) and fruit juices that contain caffeine or other methylxanthines starting two days before each administration and lasting until the last blood sample for that period is drawn. Grapefruit products should not be consumed starting seven days before the first dose is administered and lasting until the last blood sample is drawn. No food and beverages except water will be consumed starting the evening before the drug is administered, i.e. 21:00 on the evening of hospitalization and lasting until breakfast and thereafter until the lunchtime (approximately 4 hours after drug administration) in each study period. No vigorous physical activity is allowed starting two days before the initial screening tests and lasting until the last laboratory test in the final check up is performed.

Dinner on the day before drug application will be served no later than 21:00. The standardised high fat and high calorie breakfast (2 boiled eggs, 100 grams of sausage, 2 slices of toast with 10 g butter, 113 grams of hash brown potatoes with 10 g butter, 240 millilitre of whole

| Subject's paraph | | CONFIDENTIAL | | Page 1/4 |
|------------------|------------------|------------------|----------|----------|
| | Subject's paraph | | | |
| | | Subject's paraph | <u> </u> | |

**Study Code:** NOV2019/01864 **NCT04639869 Date:** 13.05.2019 **Version:** 1.0

*milk*) will be served approximately 30 minutes before the drug is administered. A typical lunch will be served approximately 4 hours after the drug is administered and a typical dinner will be served approximately 10 hours after the drug is administered. You will be fast at least 10 hours before the breakfast. The total amount of water to be consumed on the day of drug administration is maximum 1.5 litters and water consumption will begin 1 hour after the administration of the drug.

A test drug or reference drug consisting of one tablet each will be taken with 240 mL of water -as a whole in sitting position and this will be followed by mouth check. You will not be allowed to lie on your back (except sitting or walking) during **2 hours** after the drug is given. The drug will be administered approximately at 08:00-09:00 a.m.

Blood samples for drug analysis (5 mL at most each time, only in Period I; at pre-dose ( $t_0$ ) the blood sample amount will be 12 mL) will be drawn at the following times in each study period: before the drug is administered, and then 10., 20., 30., 40., 50. minutes and 1,  $1^{1/3}$ ,  $1^{2/3}$ , 2,  $2^{1/3}$ ,  $2^{2/3}$ , 3,  $3^{1/2}$ , 4, 6, 8, 10. hours after the drug is administered. Blood samples will be drawn using a catheter during the time period passed at the Clinic. The total volume of blood to be drawn during the entire study is expected to be approximately 419 mL, including blood samples for initial and final laboratory controls and the heparinised discarded blood at determined blood sampling points each of approximately 0.5 mL. An amount of blood loss could provoke; dizziness, faintness, sweating, thirst, weak and rapid pulse, rapid respiration, orthostatic hypotension and eventual decrease in some laboratory parameters such as hemoglobin and hematocrit. Having in mind that the blood loss in the present trial will take place over a period of several weeks, the risk for the volunteers to experience one of the upper side effects is relatively low.

The collected blood samples will be transferred to NOVAGENIX Bioanalytical Drug R&D Centre in Ankara-Turkey to determine the level of drug in blood. These samples will be used to only for this study and in accordance with study objectives and any remaining material will be destroyed.

You can decide at any time whether your samples can be used for the analysis of determine the level of drug in blood or should be destroyed. If you decide that your blood samples shall not be subjected to analysis, you will have to inform the investigator about your decision in a written form.

However, the samples can be stored for monitoring, inspection and audit activities of the relevant health authorities for the aim of verifying the information on clinical studies.

Samples can not be used as a source of commercial gain in any way. However, intellectual property and patent rights are exempted from this condition.

On admission to the clinic (hospitalization day in study) the luggage of all volunteers will be checked for not allowed items (food, beverages, cigarettes, chewing-gum, and any drugs). A security service personnel or clinical personnel will perform a security check on your body and on your luggage by a hand on admission to the clinic and before the start of hospitalization.

To monitor your compliance with the study, all the rooms and the corridors are being observed continuously by video cameras during the time in the clinic. All the records will be kept for 2 months after completion of the clinical period, and all records will be deleted at the end of this period.

## Side effects:

The adverse events, considered to be at least possibly related to treatment, are listed below by body system, organ class, and absolute frequency. Frequencies are defined as very common ( $\geq 1/10$ ), common ( $\geq 1/100$ ) to < 1/10), uncommon ( $\geq 1/1,000$ ) to < 1/10,000 to < 1/10,000), and very rare (< 1/10,000).

Undesirable effects in patients receiving phenyramidol are:

| 1 81 7 | |
|-------------------------------------------------------|------|
| System Organ Class | |
| Immune system disorders | |
| Hypersensitivity, pruritus, skin rash, exanthem | rare |
| Nervous system disorders | |
| Sleep disorders, sedation, dizziness, drowsiness rare | |
| Gastrointestinal disorders | |
| Nausea, vomiting, abdominal fullness | rare |
| General disorders and administration site conditions | |
| Tongue burn | rare |

(Also, a verbal explanation will be made about the unexpected side effects by the investigator.)

Please ask the informing physician about any terms you do not understand. If any side effect will occur, report to the study investigator immediately. You can ask additional questions any time during the trial about additional information not provided in this form. Investigator and authorised personnel have to be reachable 7/24 during the entire clinical study (see the phone number given in the first page).

As with all prescription drugs, other unpredictable side effects or life-threatening events can occur in addition to the above mentioned side effects. *Do not drive or operate machine on medication day.* 

Your participation of this study will be finished after the last blood sampling at  $10^{th}$  hours for pharmacokinetic purpose in the last period and the following post-study examination and laboratory tests and /or in the cases of the drop-out or occurring a serious adverse event.

Because of participating the clinical phase of the study, a payment will be done to you with a receipt/voucher or a signed minute for the loss of your working days and the some private expenditures (e.g. transportation, communication, meal, accommodation etc.). Except these, you will not have any payment for the use of blood samples obtained from clinical study or other purposes. If you violate the procedures of the study or of your own health protection, you may be withdrawn from the study before its completion or the amount of the money which will be paid to you may reduced.

**Study Code:** NOV2019/01864 NCT04639869 **Date:** 13.05.2019 **Version:** 1.0

## **Data Protection:**

Only the birth dates and initial letters of subject names will be used as identity markers in study records. Your identity will be kept confidential. Study records will only be used for scientific purposes and will be delivered to the sponsor of this study. To ensure a fair study in accordance with the rules, the authorized study monitors of the drug firm (Pharmactive İlaç San.ve Tic. A.Ş.) or the Contract Research Organisation (Novagenix), inspectors, ethics committees, and legal authorities are permitted to access your medical records. Individuals working with the study have been specially trained in this area and must adhere to occupational guidelines. They can only be given access to your personal data not including your name.

The privacy of your records will always be respected. The data protection law will be followed.

You can withdraw from the study without explanation and without risking clinical treatment that might be needed in the future. Your signature under the informed consent form does not entitle you to complete the study.

All subjects participating in this study are insured. By mutual agreement between the clinical study sponsor (Pharmactive İlaç San.ve Tic. A.Ş.) and the principal investigator, NOVAGENIX insured all participants for the cases of study-related loss of function or cases, where hospitalization or surgical intervention is required, death, or permanent disability due to this study. In case of your request a copy of the insurance policy will be given to you by investigator.

The insurer is responsible for health-related problems that may occur only under the following conditions:

- 1. Health-related issues that occur due to the treatment and/or administration of drugs with the decision and approval of the conducting physician during the research,
- 2. Any problem that may occur regarding your health due to the clinical study is immediately reported to your investigating physician and insurer by you or your relatives.

| Subject's paraph | | |
|------------------|------------|----|
| | CONFIDENTI | ΑL |

| tudy Code: NOV2019/01864 | NC104639869 | | Date: 13.05.2019<br>Version: 1.0 |
|---|---|---|---|
| Screening Number: | ) mg Film Tablet, <i>Pharmactive</i> | | (C13,011) |
| I,, agree to take part voluntarily in the above research conducted by NOVAGENIX Bioanalytical Drug R&D Centre (Contract Research Organisation) on behalf of Pharmactive İlaç San.ve Tic. A.Ş. (Sponsor) of my own free will. I have been informed about the structure of the study, its possible duration, risks and about my responsibilities by the physician whose name is given below. I have read and understood the above explanations. Physician who is responsible for informed have advised me about possible disorders and side effects. I have also read the informing document about all aspects and details of the study. Finally, I have understood and accepted all the information, explanations, and recommendations provided. | | | |
| | | the treatments and drugs I received nonths and the drug treatments I am I | d in the last three months and all the planning to take. |
| I promise to report any deterioration of my well being or my health, as well as the occurrence of any unexpected/unusual symptoms to the researchers immediately, to work in collaboration with the researchers, and to follow the instructions provided during the study. If I violate the rules, my participation to the clinical trial will be ended by the investigator(s). I have given explicit information about the previous studies in which I participated. I have been told that this research is reviewed and approved by an ethics committee. I was also told that I can ask any further questions I might have to those individuals. | | | |
| I understand that I am free to w | ithdraw from the study anytir | ne, without giving any explanation | ı <b>.</b> |
| | | | not be of direct help to my health and I de or if I do not follow the instructions |
| I promise not to behave in any wa<br>any information that might affect | | | at I will be notified immediately in case |
| I am not stipulating any restrictions for the use of study results. I accept that the results will be given to authorized people and corporations. I accept that the data recorded during the study will be delivered to the sponsor firm and later to health authorities. I understand and consent that study results will be evaluated by computer, keeping the identities of participants confidential. | | | |
| | | nsured. The sponsor drug firm appr<br>my health or wellbeing due to my pa | oves that the compensation fee will be rticipation in this study. |
| I accept that any damage that occurs to my health at my own fault and/or for disobeying the instructions of the researcher will not be covered by insurance. I have understood and accepted that damages will not be covered by insurance in case my health deteriorates due to any drugs or treatments I receive outside of the researcher's permission or knowledge. I have understood and accepted that the insurer can cover the damages that may occur due to drugs used during and for the purposes of the study, the applied procedures, or another medical treatment administration carried out by the consent of the conducting physician. | | | |
| The maximum compensation fee accepted. | to be paid in such a situation is | s up to the amount mentioned in the | insurance policy in case the liability is |
| I know that some private insurance companies accept participating in medical studies as an issue to be reported in insurance claim demands and I will check if my participation in the study will affect current policies in case of such an insurance claim demand or application for renewal. | | | |
| I or my relatives will notify the insurer and the study doctors in case any deterioration occurs in my health. I have been informed about this clinical study by verbal and by Volunteer Informed Consent Form document from an authorized medical doctor who is in the clinical study team. Also, I have read and understood this informed subject consent and study-related subject information form and accepted with my own free will, signed, and received one sample of it. | | | |
| Subject's: | | | |
| NAME | | | |
| DATE OF BIRTH | | | |
| SIGNATURE | | | |
| DATE | | | |
| As the responsible physician, I am convinced that the subject understood all the written and verbal explanations provided, read and understood the given information, and agreed to participate in the study of his/her own free will. | | | |
| <b>Doctor Who Is Responsible For</b> | Informed: | | |
| NAME | | | |
| SIGNATURE | | | |
| DATE | | | |
| This Informed Consent Form includes 4 pages. | | | |
| Subject's nameral | | | |
| Subject's paraph | | | |